CLINICAL TRIAL: NCT04875351
Title: Breast Cancer Index (BCI) Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Biotheranostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BTX-BCI-016-PRT
Record Dates: First submitted 2021-04-26; First posted 2021-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Breast Neoplasm; Invasive Breast Carcinoma; Early Stage (I, II or III) Breast Cancer; Hormone Receptor positive (HR+) Breast Cancer; Extended Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast Cancer Index (BCI) Risk of Recurrence & Extended Endocrine Benefit Testing: Female patients diagnosed with hormone receptor-positive (HR+), lymph node-negative (LN-) or lymph node-positive (LN+, with 1-3 positive nodes) early-stage invasive breast cancer, who are distant recurrence-free.
  Interventions: Diagnostic Test: Breast Cancer Index (BCI) Risk of Recurrence & Extended Endocrine Benefit Test

INTERVENTIONS:
Diagnostic Test: Breast Cancer Index (BCI) Risk of Recurrence & Extended Endocrine Benefit Test — The BCI test provides a quantitative estimate of the risk for both late (post-5 years from diagnosis) distant recurrence and of the cumulative distant recurrence risk over 10 years (0-10y) in patients treated with adjuvant endocrine therapy (LN- patients) or adjuvant chemoendocrine therapy (LN+ patients), and prediction of the likelihood of benefit from extended (>5 year) endocrine therapy.
  Other Names: Breast Cancer Index (BCI) Test

SUMMARY:
The purpose of the Breast Cancer Index (BCI) Registry study is to conduct a large scale, population-based prospective registry to evaluate long-term clinical outcome, clinical impact, medication adherence and quality of life in hormone receptor positive (HR+) early-stage breast cancer patients receiving BCI testing as part of routine clinical care to inform extended endocrine therapy.

DETAILED DESCRIPTION:
The BCI Registry is designed as a large-scale data registry and biospecimen repository to evaluate the clinical outcome of hormone receptor positive (HR+) early-stage breast cancer patients completing primary adjuvant endocrine therapy and are considering extended endocrine treatment. The impact of BCI test results on extended endocrine therapy decision-making and clinical use patterns will be characterized. Extended endocrine therapy-specific medication adherence will be assessed annually. Primary tumor tissue will be collected for scientific research purposes including molecular profiling and for correlative studies. The sample size will consist of approximately 3,000 subjects across 30-50 sites in the United States.

The BCI registry will recruit patients with HR+ stage I to III breast cancer following an initial 4-7 years of adjuvant endocrine therapy that will have BCI testing performed as part of routine clinical care and meet the inclusion/exclusion criteria. After signing the informed consent form (ICF) during screening, physicians and patients will complete the pre-test Decision Impact Questionnaire. Upon ordering BCI by the treating physician, primary tumor tissue obtained from the patient during previous breast-conserving surgery or mastectomy will be requested by Biotheranostics to perform BCI testing at Biotheranostics' CLIA certified and CAP accredited clinical laboratory in San Diego, CA. Following BCI testing, the physician will share and discuss the BCI results with their patients and recommend to either stop or extend endocrine therapy for an additional 5 years. The impact of the BCI test results on extended endocrine therapy decision-making will be assessed using the post-test Decision Impact Questionnaire, which will be completed by both physicians and patients. In addition, medication adherence will be evaluated in patients that are recommended for or elect to continue treatment to complete 10 years of adjuvant endocrine therapy.

BCI reports both a prognostic and predictive result and has been shown to significantly stratify patients based on the risk of late distant recurrence as well as to predict the likelihood of benefit from endocrine therapy in multiple prospective-retrospective studies within randomized controlled trial cohorts. The BCI registry study will determine the long-term outcome and BCI test performance to add prospective validation for the prognostic and predictive capabilities of BCI. In this context, the impact of BCI test results on treatment decision-making and subsequently prescribed treatments will be characterized.

Analysis of BCI test performance with long-term outcome will be performed by Kaplan-Meier analysis with log-rank test to assess the statistical significance of the risk stratification by BCI risk groups. Cox proportional hazards regression will be used to derive the hazard ratios (HR) and the associated 95% confidence intervals for the comparison of BCI risk groups. Univariate and multivariate analysis adjusting for clinical factors such as age, tumor size, grade, and treatment background (adjuvant endocrine therapy and chemotherapy) will be conducted. Descriptive statistics will be used to evaluate the decision-impact and medication adherence scores of patients enrolled in the study.

Each participating site will maintain appropriate medical and research records for this trial, in compliance with Section 4.9 of the ICH E6 GCP, and regulatory and institutional requirements for the protection of confidentiality of subjects. As part of participating in a Biotheranostics-sponsored study, each site will permit authorized representatives of the sponsor and regulatory agencies to examine clinical records for the purposes of quality assurance reviews, audits and evaluation of the study progress. The clinical trial manager will be in regular contact with the site research leader to check on progress and address any queries that they may have. Sites may be suspended from participating in the registry in the event of serious and persistent non-compliance with the protocol and/or Good Clinical Practice. Any major problems identified will be reported to the Trial Management Team and if necessary, the relevant regulatory bodies.

ELIGIBILITY:
Inclusion Criteria:

* Early stage (I, II or III) female breast cancer patients, who have completed 4-7 years of primary adjuvant endocrine therapy
* Patient was diagnosed with invasive breast carcinoma (ductal, lobular, or mixed ductal/lobular).
* The primary tumor was hormone receptor positive (HR+), i.e. estrogen receptor-positive and/or progesterone receptor-positive.
* The primary tumor was HER2 negative or positive and node-negative or node-positive with 1-3 positive lymph nodes.
* Subject has pre-treatment breast tumor tissue [formalin fixed and paraffin embedded (FFPE)] from a previous breast-conserving surgery, mastectomy or core needle biopsy available for testing by the Sponsor.

Exclusion Criteria:

* Patient has distant metastatic disease (M1).
* Patient was diagnosed with metaplastic breast cancer, carcinosarcoma, sarcoma, neuroendocrine carcinoma, adenoid cystic carcinoma, or phyllodes tumor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will include patients with stage I-III HR+ breast cancer that have signed an informed consent. Patients seen within a physician practice participating in the registry are potential candidates after meeting eligibility criteria requirements.
Sampling Method: Non-Probability Sample
Enrollment: 3465 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To determine BCI test performance by evaluating the long-term outcome of BCI risk groups over the follow-up period. | 5 Years
To determine medication adherence in patients undergoing extended endocrine therapy. | 5 Years
  Patients will be asked to complete a Medication Adherence Questionnaire during routine follow-up visits. Medication adherence scores over time will be evaluated in patients that are recommended for or elect to continue treatment to complete 10 years of adjuvant endocrine therapy.

SECONDARY OUTCOMES:
To prospectively assess the impact of BCI on extended endocrine therapy decision-making. | 5 Years
  The impact of the BCI test results on extended endocrine therapy decision making will be measured using pre- and post-test Decision Impact Questionnaires, which will be completed by both physicians and patients.
To correlate BCI results with molecular tumor profiles in early stage breast cancer. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A O'Shaughnessy, MD, Principal Investigator — US Oncology Network; Kai Treuner, PhD, Study Director — Biotheranostics, Inc.; Amanda KL Anderson, PhD, Study Director — Biotheranostics, Inc.
Locations (103):
- United States (103):
  - Southern Cancer Center, P.C. - Daphne, Daphne, Alabama
  - Southern Cancer Center, PC - Mobile Infirmary, Mobile, Alabama
  - Southern Cancer Center, PC - Providence Hospital, Mobile, Alabama
  - Southern Cancer Center, PC - Springhill Medical Center, Mobile, Alabama
  - Arizona Oncology Associates, PC - Glendale - Saguaro Cancer Center, Glendale, Arizona
  - Arizona Oncology Associates, PC - Goodyear, Goodyear, Arizona
  - Arizona Oncology Associates, PC - Phoenix - Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Oncology Associates, PC - Phoenix - Deer Valley, Phoenix, Arizona
  - Arizona Oncology Associates, PC - Scottsdale, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - East Valley Cancer Center, Tempe, Arizona
  - Sansum Clinic - Ridley-Tree Cancer Center, Santa Barbara, California
  - Sansum Clinic - Ridley-Tree Cancer Center (Solvang), Solvang, California
  - Rocky Mountain Cancer Center - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Center - Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Center - Centennial, Centennial, Colorado
  - Rocky Mountain Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Rocky Mountain Cancer Center - Denver Midtown, Denver, Colorado
  - Rocky Mountain Cancer Center - Denver, Denver, Colorado
  - Rocky Mountain Cancer Center - Swedish Medical Center, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Center - Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Center - Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Center - Longmont, Longmont, Colorado
  - Rocky Mountain Cancer Center - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Center - Thornton, Thornton, Colorado
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Illinois Cancer Specialists - Arlington Heights, Arlington Heights, Illinois
  - Affiliated Oncologists, LLC, Chicago Ridge, Illinois
  - Illinois Cancer Specialists - Niles, Niles, Illinois
  - Maryland Oncology Hematology, P.A. - Bethesda, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A. - Brandywine, Brandywine, Maryland
  - Maryland Oncology Hematology, P.A. - Clinton, Clinton, Maryland
  - Maryland Oncology Hematology, P.A. - Columbia, Columbia, Maryland
  - Maryland Oncology Hematology, P.A. - Frederick, Frederick, Maryland
  - Maryland Oncology Hematology, P.A. - Lanham, Lanham, Maryland
  - Maryland Oncology Hematology, P.A. - Rockville - Aquilino Cancer Center, Rockville, Maryland
  - Maryland Oncology Hematology, P.A. - Silver Spring - White Oak Cancer Center, Silver Spring, Maryland
  - New York Oncology Hematology, P.C. - Albany Cancer Center, Albany, New York
  - New York Oncology Hematology, P.C. - Albany Medical Center, Albany, New York
  - Broome Oncology, LLC - Binghamton, Binghamton, New York
  - New York Oncology Hematology, P.C. - Clifton Park Cancer Center, Clifton Park, New York
  - Broome Oncology, LLC - Johnson City, Johnson City, New York
  - Alliance Cancer Specialists, PC, Bensalem, Pennsylvania
  - Consultants In Medical Oncology and Hematology, P.C., Broomall, Pennsylvania
  - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - Alliance Cancer Specialists, PC, Langhorne, Pennsylvania
  - Alliance Cancer Specialists, PC, Philadelphia, Pennsylvania
  - Alliance Cancer Specialists, PC, Sellersville, Pennsylvania
  - Alliance Cancer Specialists, PC, Wynnewood, Pennsylvania
  - Texas Oncology - Abilene, Abilene, Texas
  - Texas Oncology - Allen, Allen, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology - DFWW, Arlington, Texas
  - Texas Oncology - Beaumont, Beaumont, Texas
  - Texas Oncology - Beaumont Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology - DFWW, Bedford, Texas
  - Texas Oncology - Carrollton, Carrollton, Texas
  - Texas Oncology - DFWW, Dallas, Texas
  - Texas Oncology - Medical City Dallas, Dallas, Texas
  - Texas Oncology - Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Denison, Denison, Texas
  - Texas Oncology - Denton, Denton, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Gateway, El Paso, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Joe Battle, El Paso, Texas
  - Texas Oncology - Flower Mound, Flower Mound, Texas
  - Texas Oncology - DFWW, Grapevine, Texas
  - Texas Oncology - Harlingen, Harlingen, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology - Willowbrook, Houston, Texas
  - Texas Oncology - Northeast Texas, Longview, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology - Midland, Midland, Texas
  - Texas Oncology - New Braunfels, New Braunfels, Texas
  - Texas Oncology - Odessa, Odessa, Texas
  - Texas Oncology - Northeast Texas, Palestine, Texas
  - Texas Oncology - Northeast Texas, Paris, Texas
  - Texas Oncology - Plano West, Plano, Texas
  - Texas Oncology - San Antonio Downtown, San Antonio, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - San Antonio Stone Oak, San Antonio, Texas
  - Texas Oncology - Sugar Land, Sugar Land, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Texas Oncology - Austin, Waco, Texas
  - Texas Oncology - Horizon Circle, Waco, Texas
  - Texas Oncology - Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology - Weslaco, Weslaco, Texas
  - Texas Oncology - Wichita Falls, Wichita Falls, Texas
  - Virginia Cancer Specialists, PC - Alexandria, Alexandria, Virginia
  - Virginia Cancer Specialists, PC - Arlington, Arlington, Virginia
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Cancer Specialists, PC - Fairfax, Fairfax, Virginia
  - Virginia Cancer Specialists, PC - Gainesville, Gainesville, Virginia
  - Virginia Cancer Specialists, PC - Loudoun, Leesburg, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Oncology Associates, Williamsburg, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noordhoek I, Treuner K, Putter H, Zhang Y, Wong J, Meershoek-Klein Kranenbarg E, Duijm-de Carpentier M, van de Velde CJH, Schnabel CA, Liefers GJ. Breast Cancer Index Predicts Extended Endocrine Benefit to Individualize Selection of Patients with HR+ Early-stage Breast Cancer for 10 Years of Endocrine Therapy. Clin Cancer Res. 2021 Jan 1;27(1):311-319. doi: 10.1158/1078-0432.CCR-20-2737. Epub 2020 Oct 27. PMID 33109739
- [Background] Bartlett JMS, Sgroi DC, Treuner K, Zhang Y, Ahmed I, Piper T, Salunga R, Brachtel EF, Pirrie SJ, Schnabel CA, Rea DW. Breast Cancer Index and prediction of benefit from extended endocrine therapy in breast cancer patients treated in the Adjuvant Tamoxifen-To Offer More? (aTTom) trial. Ann Oncol. 2019 Nov 1;30(11):1776-1783. doi: 10.1093/annonc/mdz289. PMID 31504126
- [Background] Zhang Y, Schnabel CA, Schroeder BE, Jerevall PL, Jankowitz RC, Fornander T, Stal O, Brufsky AM, Sgroi D, Erlander MG. Breast cancer index identifies early-stage estrogen receptor-positive breast cancer patients at risk for early- and late-distant recurrence. Clin Cancer Res. 2013 Aug 1;19(15):4196-205. doi: 10.1158/1078-0432.CCR-13-0804. Epub 2013 Jun 11. PMID 23757354
- [Background] Sgroi DC, Sestak I, Cuzick J, Zhang Y, Schnabel CA, Schroeder B, Erlander MG, Dunbier A, Sidhu K, Lopez-Knowles E, Goss PE, Dowsett M. Prediction of late distant recurrence in patients with oestrogen-receptor-positive breast cancer: a prospective comparison of the breast-cancer index (BCI) assay, 21-gene recurrence score, and IHC4 in the TransATAC study population. Lancet Oncol. 2013 Oct;14(11):1067-1076. doi: 10.1016/S1470-2045(13)70387-5. Epub 2013 Sep 12. PMID 24035531
- [Background] Sgroi DC, Carney E, Zarrella E, Steffel L, Binns SN, Finkelstein DM, Szymonifka J, Bhan AK, Shepherd LE, Zhang Y, Schnabel CA, Erlander MG, Ingle JN, Porter P, Muss HB, Pritchard KI, Tu D, Rimm DL, Goss PE. Prediction of late disease recurrence and extended adjuvant letrozole benefit by the HOXB13/IL17BR biomarker. J Natl Cancer Inst. 2013 Jul 17;105(14):1036-42. doi: 10.1093/jnci/djt146. Epub 2013 Jun 28. PMID 23812955